CLINICAL TRIAL: NCT02034773
Title: A Phase 1, Three-part Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple Doses of CC-220 and to Evaluate the Relative Bioavailability of a Formulated CC-220 Capsule in Healthy Subjects
Brief Title: 3-part Study to Evaluate Safety, Tolerability, Pharmacokinetics & Pharmacodynamics of Multiple Doses of CC-220 and Relative Bioavailability of a Formulated CC-220 Capsule
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene Corporation (Industry)
Responsible Party: Sponsor
Organization: Celgene (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: CC-220-CP-002
Record Dates: First submitted 2014-01-10; First posted 2014-01-13 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2014-01

CONDITIONS: Healthy Volunteers
Keywords: Safety, Pharmacokinetics, Pharmacodynamics, Healthy Subjects
MeSH Terms: interventions — iberdomide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- CC-220 0.3mg x 14 days (Experimental)
  Interventions: Drug: CC-220
- CC-220 1mg x 28 days (Experimental)
  Interventions: Drug: CC-220
- CC-220 0.3mg x 28 days (Experimental)
  Interventions: Drug: CC-220
- CC-220 1mg x a total of 14 days (Experimental)
  Interventions: Drug: CC-220
- Placebo (Experimental)
  Interventions: Drug: Placebo
- CC-220 0.3mg (once every 3 days for 14 days) (Experimental)
  Interventions: Drug: CC-220
- CC-220 1mg (once every 7 days for 28 days) (Experimental)
  Interventions: Drug: CC-220
- CC-220 1mg (formulated and reference capsules) (Experimental)
  Interventions: Drug: CC-220

INTERVENTIONS:
Drug: CC-220 — CC-220 0.3mg will be administered once daily for 14 days
  Arms: CC-220 0.3mg x 14 days
Drug: CC-220 — CC-220 1mg will be administered once daily for 28 days + 1 dose of tetanus toxoid vaccination and 1 dose of pneumococcal vaccination
  Arms: CC-220 1mg x 28 days
Drug: CC-220 — CC-220 0.3mg will be administered once daily for 28 days
  Arms: CC-220 0.3mg x 28 days
Drug: CC-220 — CC-220 1mg will be administered once daily for 7 days on 2 separate occasions, with a 7-day washout in between, for a total of 14 days of dosing
  Arms: CC-220 1mg x a total of 14 days
Drug: Placebo — Placebo will be administered once daily for up to 28 days
  Arms: Placebo
Drug: CC-220 — CC-220 0.3mg will be administered every 3 days for 14 days (5 total doses)
  Arms: CC-220 0.3mg (once every 3 days for 14 days)
Drug: CC-220 — CC-220 1mg (once every 7 days for 28 days)
  Arms: CC-220 1mg (once every 7 days for 28 days)
Drug: CC-220 — CC-220 1mg will be administered as a single dose in each of 2 study periods; once as a formulated capsule and once as two reference capsules
  Arms: CC-220 1mg (formulated and reference capsules)

SUMMARY:
To evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of multiple doses of CC-220 in healthy subjects and to evaluate the relative bioavailability of a formulated CC-220 capsule

DETAILED DESCRIPTION:
This is a 3-part study to be conducted at a single study center. Part 1 is a randomized, double-blind, placebo-controlled, ascending-dose study. During the course of Part 1, each subject will participate in a screening phase, a baseline phase, a treatment phase and a follow up visit. There will be a total of 4 cohorts, each of which consists of a different dose level and/or dosing duration, with 8 or 9 subjects per cohort. In each cohort, 6 subjects will receive a dose of CC-220 and the remaining subjects will receive placebo depending on the randomization schedule. In 2 of the cohorts, study drug will be administered once daily for a total of 14 days. In the other 2 cohorts, study drug will be administered once daily for 28 days. In one of the 28-day dosing cohorts, 2 vaccinations (tetanus toxoid adsorbed and pneumococcal vaccinations) will also be administered on Day 14 of the 28-day dosing period to help characterize the effect of CC-220 on antibody responses. Part 2 is a randomized, double-blind, placebo-controlled, parallel-group study to explore the effects of an alternative dosing schedule on the pharmacodynamics of CC-220. During the course of Part 2, each subject will participate in a screening phase, a baseline phase, a treatment phase and a follow up visit. There will be a total of 2 cohorts, each of which consists of a different dose level, with 9 subjects per cohort. In each cohort, 6 subjects will receive a dose of CC-220 and 3 subjects will receive placebo depending on the randomization schedule. The dosing frequency will be either once every 3 days for 14 days or once every 7 days for 28 days. Part 3 is a randomized, open-label, two-period, two-way crossover study to evaluate the relative bioavailability of one CC-220 formulated capsule, relative to two reference capsules, following a single oral dose of CC-220. During the course of Part 3, each subject will participate in a screening phase, a baseline phase, a treatment phase consisting of 2 periods, and a follow up visit. There will be one cohort consisting of a total of 12 subjects. In each study period, approximately 6 subjects will receive a single dose of CC-220 as one formulated capsule (test product) and approximately 6 subjects will receive a single dose of CC-220 as two reference capsules (reference product).

ELIGIBILITY:
Inclusion Criteria:

* 1. Must understand and voluntarily sign a written informed consent document prior to any study-related procedures being performed.

  2. Must be able to communicate with the investigator, understand and comply with the requirements of the study, and agree to adhere to restrictions and examination schedules.

  3. Healthy male or female of any race between 18 to 55 years of age (inclusive) at the time of signing the informed consent document, and in good health as determined by a physical examination.

  4. For males: Agree to use barrier contraception not made of natural (animal) membrane [e.g., latex or polyurethane condoms are acceptable]) when engaging in sexual activity with a female of childbearing potential while on study medication, and for at least 28 days after the last dose of study medication.

For females: Female subjects must have been surgically sterilized (hysterectomy or bilateral oophorectomy; proper documentation required) at least 6 months before screening, or be postmenopausal (defined as 24 months without menses before screening, with an estradiol level of < 30 pg/mL and follicle-stimulating hormone level of > 40 IU/L at screening).

5. Must have a body mass index between 18 and 33 kg/m2 (inclusive). 6. Clinical laboratory tests must be within normal limits or acceptable to the investigator. Platelet count, absolute neutrophil count and absolute lymphocyte count must be above the lower limit of normal at the screening visit.

7. Subject must be afebrile, with supine systolic blood pressure: 90 to 140 mmHg, supine diastolic blood pressure: 50 to 90 mmHg, and pulse rate: 40 to 110 bpm.

8. Must have a normal or clinically-acceptable 12-lead electrocardiogram at screening. Male subjects must have a QTcF value ≤ 430 msec. Female subjects must have a QTcF value ≤ 450 msec.

9. Antitetanus immunoglobulin G titer ≥ 0.1 IU/mL to ensure prior exposure of tetanus toxoid. Note: This criterion only applies to those subjects who will be dosed once daily for 28 days.

Exclusion Criteria:

* 1. History of any clinically significant and relevant neurological, gastrointestinal, renal, hepatic, cardiovascular, psychological, pulmonary, metabolic, endocrine, hematological, allergic disease, drug allergies, or other major disorders.

  2. Any condition which places the subject at unacceptable risk if he or she were to participate in the study, or confounds the ability to interpret data from the study.

  3. Used any prescribed systemic or topical medication (including but not limited to analgesics, anesthetics, etc) within 30 days of the first dose administration, unless sponsor agreement is obtained.

  4. Used any non-prescribed systemic or topical medication (including vitamin/mineral supplements, and herbal medicines) within 14 days of the first dose administration, unless sponsor agreement is obtained.

  5. Used CYP3A inducers and inhibitors (including St. John's Wort) within 30 days of the first dose administration.

  6. Has any surgical or medical conditions possibly affecting drug absorption, distribution, metabolism and excretion, e.g., bariatric procedure. Appendectomy and cholecystectomy are acceptable.

  7. Donated blood or plasma within 8 weeks before the first dose administration to a blood bank or blood donation center.

  8. History of drug abuse (as defined by the current version of the Diagnostic and Statistical Manual) within 2 years before dosing, or positive drug screening test reflecting consumption of illicit drugs.

  9. History of alcohol abuse (as defined by the current version of the Diagnostic and Statistical Manual) within 2 years before dosing, or positive alcohol screen.

  10. Known to have serum hepatitis or known to be a carrier of hepatitis B surface antigen or hepatitis c antibody, or have a positive result to the test for human immunodeficiency virus antibodies at screening.

  11. Exposed to an investigational drug (new chemical entity) within 30 days preceding the first dose administration, or 5 half-lives of that investigational drug, if known (whichever is longer).

  12. Smoke more than 10 cigarettes per day, or the equivalent in other tobacco products (self reported).

  13. Vaccination within 30 days of dosing or plans to receive vaccination within 30 days after dosing. Systemic infection within 30 days of dosing.

  14. Tetanus vaccination within 5 years prior to the first dose administration. Note: This criterion only applies to those subjects who will be dosed once daily for 28 days.

  15. Pneumococcal vaccination within 3 years prior to the first dose administration. Note: This criterion only applies to those subjects who will be dosed once daily for 28 days.

  16. Any self-reported history of hypersensitivity to vaccinations to be administered in this study or hypersensitivity to latex. Note: This criterion only applies to those subjects who will be dosed once daily for 28 days.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2013-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Up to 7 months overall
  Number of participants with adverse events

SECONDARY OUTCOMES:
Concentrations of CC-220 and its R-enantiomer in plasma | Up to 30 days per cohort
  Blood samples will be collected at pre-specified times to determine levels of CC-220 and its R-enantiomer in plasma
Pharmacodynamic Assessmens | Up to 42 days per cohort
  Blood samples will be collected at pre-specified times for pharmacodynamic assessments
Pharmacokinetics - Cmax | Up to 30 days
  Maximum observed plasma concentration
Pharmacokinetics - tmax | Up to 30 days
  Time to Cmax
Pharmacokinetics - AUCinf | Up to 30 days
  Area under the plasma concentration-time curve from time zero extrapolated to infinity
Pharmacokinetics - AUCt | Up to 30 days
  Area under the plasma concentration-time curve from time zero to the last quantifiable concentration
Pharmacokinetics - AUCtau | Up to 30 days
  Area under the plasma concentration-time curve from time zero to tau, where tau is the dosing interval
Pharmacokinetics - t1/2,z | Up to 30 days
  Terminal-phase elimination half-life
Pharmacokinetics - CL/F | Up to 30 days
  Apparent total plasma clearance when dosed orally
Pharmacokinetics - Vz/F | Up to 30 days
  Apparent total volume of distribution when dosed orally, based on the terminal phase
Accumulation Ratio (RA) | Up to 30 days
  Accumulation Ratio for Cmax and AUCtau

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Weiss, MD, Study Director — Celgene; Debra Mandarino, MD, Principal Investigator — Covance
Locations (1):
- Covance Clinical Research Unit, Madison, Wisconsin, United States